CLINICAL TRIAL: NCT06977984
Title: Group Breathwork Intervention for Chronic Pain
Brief Title: Group Integrative Breathwork for Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500383
Record Dates: First submitted 2025-05-06; First posted 2025-05-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
Keywords: Breathwork; Chronic Pain; Integrative Breathwork Intervention; Chronic Musculoskeletal Pain; Breathing Therapy; Intervention Development
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: We will conduct multiple single-arm iterations testing and refining the group breathwork intervention prior to conducting a pilot randomized controlled trial comparing the refined version of the intervention to a waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative Breathwork Intervention (Experimental): The breathwork intervention will be delivered in groups of 2-5 participants with chronic musculoskeletal pain. A conscious connected breathing technique will be engaged in for 45-60 minutes.
  Interventions: Behavioral: Integrative Breathwork Intervention

INTERVENTIONS:
Behavioral: Integrative Breathwork Intervention — The breathwork intervention involves a sustained conscious connected breathing pattern where there is no pause between inhale and exhale. During the breathing, a participant is guided to pay attention to the strongest sensation from moment-to-moment (e.g., mindfulness of somatic sensations) and relax unnecessary effort or tension. Participants lay supine throughout the 60 minute session. The session ends with spontaneous, relaxed breathing and an opportunity to briefly share one's experience.

SUMMARY:
The aim of the proposed research is to iteratively develop, pilot test, and refine an integrative breathwork intervention that is suitable for group delivery to individuals with chronic pain. The intervention will be evaluated for feasibility, acceptability, and plausibility for clinically significant effects in people with chronic musculoskeletal pain.

DETAILED DESCRIPTION:
Multiple single-arm iterations of a group breathwork intervention will be conducted to refine and optimize the intervention and protocol. Upon completion of each iteration, quantitative and qualitative data will be gathered to identify possible modifications before proceeding with the next iteration. After achieving a satisfactory intervention, we will conduct a pilot randomized controlled trial compared to a waitlist control group. This work will provide initial evidence on the feasibility, acceptability, and plausibility of clinically significant effects of this type of multicomponent breathwork intervention for adults with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-70 years of age.
2. Chronic musculoskeletal pain lasting for at least 3 months as a symptom of axial pain (e.g., back, neck) or limb pain (e.g., shoulder, knee, hip, wrist).
3. Average pain intensity of ≥ 4/10 for the past month.
4. Access to internet with a valid email address
5. Able to lay down and stay relatively still for one hour.

Exclusion Criteria:

1. Any suspicion of a medical (orthopedic, rheumatic or neurological) disease, that can fully explain the current level of severity of pain.
2. Chronic pain possibly due to specific conditions (e.g., cancer, infection).
3. Ongoing legal action or disability claim related to chronic pain.
4. Neurological disease (e.g. Parkinson's, multiple sclerosis, epilepsy, history of seizures) or moderate or severe symptoms from a previous brain injury, including stroke and traumatic brain injury.
5. Respiratory disorder (e.g., chronic obstructive pulmonary disease) or moderate to severe asthma within the past 12 months.
6. Activity limiting heart disease including cardiovascular or peripheral arterial disease.
7. Uncontrolled hypertension (i.e. SBP/DBP of > 160/95) or orthostatic hypotension (e.g., issues with fainting).
8. Serious acute physical injuries or major surgery within the past 6 months.
9. Serious psychiatric disorder (e.g., schizophrenia, panic disorder) or mental health issues requiring hospitalization within the past 12 months or currently on antipsychotic medications.
10. History of hospitalization or treatment of substance use disorder within the past 12 months.
11. Currently undergoing curative or palliative chemotherapy or radiation.
12. Pregnant.
13. Glaucoma or detached retina.
14. Current participation or participation in the past 2 months of an interventional research study.
15. Cognitive impairment or factors that would preclude comprehension of material and/or full participation in the study.
16. Any significant comorbidities or other reasons that, in the opinion of the investigators, could interfere with the study or lead to deleterious effects for the participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability | Day 1
  Treatment acceptability and satisfaction of the breathwork intervention will be measured using several face-valid items rated on a 10-point scale (1-10) where higher scores represent greater treatment acceptability and satisfaction.
Change in Pain Intensity and Interference | Change from Baseline to 1-week follow-up, 1-month follow-up
  The Pain, Enjoyment, and General Activities (PEG-3) scale will be used to assess pain intensity and pain interference over the past week on average.

SECONDARY OUTCOMES:
Patient's Global Impressions of Change | 1-week follow-up, 1-month follow-up
  The Patient's Global Impression of Change single-item measure asks participants to describe any changes in activity limitations, symptoms, emotions, and overall quality of life, related to their pain since the beginning of the treatment. (Higher scores represent greater impressions of benefit from the intervention.)
Change in Pain Catastrophizing | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the 13-item Pain Catastrophizing Scale. (Scores range from 0-52; higher scores represent higher levels of pain catastrophizing).
Acute Treatment Effects | Day 1
  Assessed using face-valid items related to feelings and emotions immediately before and after the intervention session. Scores will be calculated by subtracting post-intervention to pre-intervention where higher scores represent greater acute subjective effects.
Change in Pain Self-Efficacy | Change from Baseline to 1-month follow-up
  Assessed using the 10-item Pain Self-Efficacy Scale. (0-6; higher scores represent higher levels of pain self-efficacy).
Change in Sleep Disturbances | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the PROMIS-Sleep Disturbance 8b scale. (1-5; higher scores represent higher levels of sleep disturbance).
Change in Sleep Related Impairment | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the PROMIS-Sleep Related Impairment 8a scale. (1-5; higher scores represent higher levels of sleep related impairment).
Change in Fatigue | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the PROMIS Fatigue-8a scale. (1-5; higher scores represent higher levels of fatigue over the past week).
Change in Whole Person Health | Change from Baseline to 1-month follow-up
  Assessed using the Whole Person Health Index. (1-5; lower scores represent better levels of self-assessed health ).
Change in Stress | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the 4-item Perceived Stress Scale. (0-4; higher scores represent higher levels of subjective stress over the past month).
Change in Anxiety | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the Generalized Anxiety Disorder-2 Questionnaire. (0-3; higher scores represent higher levels of anxiety over the past 2 weeks).
Change in Depression | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the Patient Health Questionnaire-2.(0-3; higher scores represent higher levels of depression over the past 2 weeks).
Change in Fear Avoidance Beliefs | Change from Baseline to 1-week follow-up, 1-month follow-up
  Assessed using the 5-item Fear-Avoidance Beliefs Questionnaire-physical activity subscale. (0-6; higher scores represent higher levels of physical activity-related fear-avoidance beliefs).
Change in Interoception | Change from Baseline to 1-month follow-up
  Assessed using the Multidimensional Assessment of Interoceptive Awareness-2. (0-5; higher scores represent higher levels of interoception).
Change in Multisensory Sensitivity | Change from Baseline to 1-month follow-up
  Assessed using the Multisensory Amplification Scale will be used to assess symptoms of central nervous system hypersensitivity, or central sensitization. (1-5; higher scores represent higher levels of sensory sensitivity).
Psychological Insight | 1-month follow-up
  Assessed using the Psychological Insight Questionnaire where higher scores represent greater levels of psychological insight arising from the breathwork intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided